CLINICAL TRIAL: NCT06834243
Title: Comparison of Intermittent Bolus and Continuous Infusion Pericapsular Nerve Group Block on Recovery Quality and Analgesic Consumption: a Retrospective Study
Brief Title: Comparison of Intermittent Bolus Vs. Continuous Infusion PENG Block for Postoperative Pain in Hip Surgery
Acronym: ICPENG
Status: Completed | Type: Observational
Sponsor: Onur Baran (Other)
Collaborators: Namik Kemal University School of Medicine, Tekirdag (Other)
Responsible Party: Sponsor-Investigator, Onur Baran, Asst. Prof., Namik Kemal University
Organization: Namik Kemal University (Other)
Other Study IDs: TNKU-PENG-Retro
Record Dates: First submitted 2025-02-12; First posted 2025-02-19 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Hip Surgery; Postoperative Pain Management; Pericapsular Nerve Group Block (PENG Block); Regional Anesthesia
Keywords: Hip surgery; postoperative pain; pericapsular nerve group block; analgesia
MeSH Terms: conditions — Pain, Postoperative; Agnosia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Intermittent Bolus Group: Patients in this group received intermittent bolus administration of the Pericapsular Nerve Group (PENG) Block via a catheter placed under ultrasound guidance at the end of surgery. A researcher manually administered 20 mL of 0.25% bupivacaine every 4 hours over a 24-hour period.
  * Total bupivacaine volume: 120 mL of 0.25% bupivacaine over 24 hours
  * Additional analgesia: All patients received PCA with tramadol, IV paracetamol, and rescue NSAIDs as per protocol.
  Interventions: Procedure: Intermittent Bolus PENG Block
- Continuous Infusion Group: Patients in this group received continuous infusion of the Pericapsular Nerve Group (PENG) Block via a catheter placed under ultrasound guidance at the end of surgery. A pump delivered 5 mL/hour of 0.25% bupivacaine continuously over a 24-hour period.
  * Total bupivacaine volume: 120 mL of 0.25% bupivacaine over 24 hours
  * Additional analgesia: All patients received PCA with tramadol, IV paracetamol, and rescue NSAIDs as per protocol.
  Interventions: Procedure: Continuous Infusion PENG Block

INTERVENTIONS:
Procedure: Intermittent Bolus PENG Block — Patients received intermittent bolus administration of the Pericapsular Nerve Group (PENG) Block via a catheter. A researcher manually administered 20 mL of 0.25% bupivacaine every 4 hours over a 24-hour period.
  Groups: Intermittent Bolus Group
Procedure: Continuous Infusion PENG Block — Patients received continuous infusion of the Pericapsular Nerve Group (PENG) Block via a catheter. A pump delivered 5 mL/hour of 0.25% bupivacaine continuously over a 24-hour period.
  Groups: Continuous Infusion Group

SUMMARY:
This retrospective study evaluates the effects of two different administration methods of the Pericapsular Nerve Group (PENG) Block on postoperative pain control, opioid consumption, and recovery in patients undergoing hip surgery.

All patients in the study received:

* PENG block via a catheter
* Patient-Controlled Analgesia (PCA) with tramadol
* Multimodal analgesia, including IV paracetamol and nonsteroidal anti inflammatory drugs (NSAIDs) as rescue analgesia

The study compares two groups:

1. Intermittent Bolus Group: A researcher administered 20 mL of 0.25% bupivacaine every 4 hours.
2. Continuous Infusion Group: A pump delivered 5 mL/hour of 0.25% bupivacaine continuously.

Both groups received the same total volume of local anesthetic over 24 hours. All PENG blocks were performed under ultrasound guidance at the end of surgery. This study aims to determine whether intermittent bolus or continuous infusion PENG block administration leads to better pain control, lower opioid consumption, and improved recovery outcomes.

DETAILED DESCRIPTION:
Postoperative pain management after hip surgery remains a critical factor in recovery quality, opioid consumption, and overall patient outcomes. Among regional anesthesia techniques, the PENG Block is increasingly utilized for pain control due to its ability to provide effective analgesia while minimizing systemic opioid use. However, the optimal administration method of PENG block remains unclear.

This retrospective cohort study evaluates the effectiveness of two different PENG block administration techniques in patients undergoing hip surgery:

1. Intermittent Bolus Group: A researcher manually administered 20 mL of 0.25% bupivacaine every 4 hours via a catheter placed under ultrasound guidance at the end of surgery.
2. Continuous Infusion Group: A pump delivered 5 mL/hour of 0.25% bupivacaine continuously via a catheter placed under ultrasound guidance at the end of surgery.

Total local anesthetic volume over 24 hours was equal in both groups.

Study Objectives:

The primary objective is to compare intermittent bolus vs. continuous infusion PENG block administration in terms of:

* Postoperative pain control (Visual Analog Scale) (VAS scores)
* Total opioid consumption (morphine equivalent)
* Time to first rescue analgesia
* Quality of recovery (QoR-15 at 24 hours postoperative)

Secondary outcomes include:

* Postoperative nausea and vomiting (PONV)
* Incidence of complications (hematoma, infection, nerve injury)

This study aims to provide evidence on whether intermittent bolus or continuous infusion leads to better pain relief, reduced opioid consumption, and improved recovery in hip surgery patients.

ELIGIBILITY:
Inclusion Criteria

Participants must meet all of the following criteria to be included in the study:

1. Patients who underwent hip surgery between November 15, 2023 - November 15, 2024.
2. Patients who received Pericapsular Nerve Group (PENG) Block via a catheter for postoperative analgesia.
3. Patients who received Patient-Controlled Analgesia (PCA) with tramadol.
4. Patients aged 18 to 65 years.
5. ASA I - III classification.
6. BMI ≤ 35 kg/m². Exclusion Criteria

Participants who meet any of the following criteria will be excluded from the study:

1. Patients who received analgesia with techniques other than PENG block.
2. Patients with incomplete or missing medical records.
3. Patients with a psychiatric illness diagnosis that may interfere with pain perception or reporting.
4. Patients with coagulation disorders (e.g., INR >1.5, thrombocytopenia).
5. Patients with hepatic or renal failure (Creatinine clearance <30 mL/min or AST/ALT >3x normal).
6. Patients with chronic opioid use before surgery.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study includes adult patients (ages 18-65) who underwent hip surgery at Tekirdağ Namık Kemal University Hospital between November 15, 2023, and November 15, 2024. All patients received Pericapsular Nerve Group (PENG) Block via a catheter for postoperative pain management, along with multimodal analgesia including tramadol PCA, IV paracetamol, and rescue NSAIDs. The study compares two PENG block administration techniques: intermittent bolus versus continuous infusion.
Sampling Method: Non-Probability Sample
Enrollment: 82 (Actual)
Dates: Start 2023-11-15 (Actual); Primary Completion 2024-11-15 (Actual); Study Completion 2024-11-15 (Actual)

PRIMARY OUTCOMES:
Total Postoperative Opioid Consumption | From 0 hours (postoperatively) to 24 hours postoperatively, assessed at 0, 2, 6, 12, and 24 hours.
  Total opioid consumption (including PCA tramadol) will be recorded and converted into morphine milligram equivalents (MME) for comparison between groups.
Quality of Recovery (QoR-15 Score) | Assessed at 24 hours postoperatively.
  The Quality of Recovery-15 (QoR-15) questionnaire will be used to assess the patient's postoperative recovery quality, including physical and emotional well-being. The QoR-15 is a validated tool that measures postoperative recovery across five domains: physical comfort, emotional state, psychological support, physical independence, and pain.
  Scale Range: 0 to 150 Interpretation: Higher scores indicate better recovery quality. Time Frame: Assessed at 24 hours postoperatively.
Time to First Rescue Analgesia | From the end of surgery until the first administration of rescue analgesia, assessed up to 24 hours postoperatively.
  The time from surgery completion to the first NSAID rescue analgesia administration (ketorolac or dexketoprofen) will be recorded.
Postoperative Pain Scores (VAS) | From 0 hours (postoperatively) to 24 hours postoperatively, assessed at 0, 2, 6, 12, and 24 hours.
  Postoperative pain levels will be assessed using the Visual Analog Scale (VAS, 0-10) where:
  * 0 = No pain
  * 10 = Worst possible pain
  * Higher scores indicate worse pain levels.

SECONDARY OUTCOMES:
Postoperative Nausea and Vomiting (PONV) Incidence | From 0 hours (postoperatively) to 24 hours postoperatively.
  Incidence of postoperative nausea and vomiting (PONV) will be recorded based on medical chart reviews and antiemetic administration (ondansetron IV use).
Incidence of Complications | From 0 hours (postoperatively) to 24 hours postoperatively.
  Any adverse events (hematoma, infection, nerve injury, hemodynamic instability, etc.) will be documented from patient records.

CONTACTS AND LOCATIONS:
Overall Officials: Cavidan Arar, Prof. Dr., Study Chair — Medical Faculty of Tekirdağ Namık Kemal University
Locations (1):
- Tekirdağ Namık Kemal University Research Hospital, Tekirdağ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to ethical considerations and institutional privacy regulations. Only de-identified, aggregated results will be published in scientific journals and conferences."

REFERENCES:
- [Background] Huda AU, Ghafoor H. The Use of Pericapsular Nerve Group (PENG) Block in Hip Surgeries Is Associated With a Reduction in Opioid Consumption, Less Motor Block, and Better Patient Satisfaction: A Meta-Analysis. Cureus. 2022 Sep 6;14(9):e28872. doi: 10.7759/cureus.28872. eCollection 2022 Sep. PMID 36105907
- [Background] Kukreja P, Uppal V, Kofskey AM, Feinstein J, Northern T, Davis C, Morgan CJ, Kalagara H. Quality of recovery after pericapsular nerve group (PENG) block for primary total hip arthroplasty under spinal anaesthesia: a randomised controlled observer-blinded trial. Br J Anaesth. 2023 Jun;130(6):773-779. doi: 10.1016/j.bja.2023.02.017. Epub 2023 Mar 22. PMID 36964012